CLINICAL TRIAL: NCT02374450
Title: A Prospective Study to Estimate the Incidence of Diseases Specified as Adverse Events of Special Interest, of Other Adverse Events Leading to Hospitalisation or Death, and of Meningitis in Infants and Young Children in Sub-Saharan Africa Prior to Implementation of the RTS,S/AS01E Candidate Vaccine
Brief Title: A Surveillance Study of Diseases Specified as Adverse Events of Special Interest, of Other Adverse Events Leading to Hospitalisation or Death, and of Meningitis in Children in Africa Prior to Implementation of the RTS,S/AS01E Candidate Vaccine
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PATH (Other); Agence de Médecine Préventive, France (Other); Réseau en Afrique Francophone pour la Télémédecine, (Other); Iqvia Pty Ltd (Industry); Parexel (Industry); Clinical Laboratory Services (Other)
Responsible Party: Sponsor
Other Study IDs: 115055
Record Dates: First submitted 2015-01-12; First posted 2015-02-27 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Malaria
Keywords: Malaria; Surveillance study; Adverse Events of Specific Interest (AESI); Children; Infants; Adverse events (AE) leading to hospitalisation or death; Meningitis; Epidemiology; Africa
MeSH Terms: conditions — Malaria; Death; Meningitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Active surveillance 6-12 weeks: Children were identified at the first administration of Diphtheria-tetanus-whole- cell pertussis-hepatitis B- Haemophilus influenza type b pentavalent (DTP/HepB/Hib) vaccine (usually given at 6weeks of age) and home visits were conducted according to DTP/HepB/Hib vaccine schedule.
  Interventions: Procedure: Blood collection
- Active surveillance 5-17 months: Children who were either identified at the first administration of the DTP/HepB/Hib vaccine (usually given at 6 weeks of age), with home visits scheduled from 5 months of age onwards or identified at first encounter with the study staff, with home visits started within one week of the first encounter with study staff.
  Interventions: Procedure: Blood collection
- Enhanced hospitalization surveillance: All children under the age of 5 years within the study areas, who were not already enrolled in active surveillance were eligible for enrolment in enhanced hospitalization surveillance during any hospitalizations throughout the entire study period.
  Interventions: Procedure: Blood collection

INTERVENTIONS:
Procedure: Blood collection — For all hospitalised children suspected of having an AESI or meningitis, a sample of 5 ml of whole blood was collected and the serum was stored.

SUMMARY:
The purpose of this pre-licensure cohort study was to estimate the incidence of adverse events of special interest (AESI), other adverse events (AE) leading to hospitalisation or death, meningitis and malaria in sub-Saharan African children under 5 years of age. The outcomes of this study provide the baseline data for the post-licensure EPI-MALARIA-003 (115056) study that evaluated the safety, effectiveness and impact of the RTS,S/AS01E vaccine.

An interim analysis was performed on a sub-group of study participants enrolled in active surveillance from sites where the vaccine was implemented, having 6 months of follow-up after the administration of dose 3 of DTP/HepB/Hib vaccine (6-12 weeks group), or 6 months after Visit 3 (mimicking the RTS,S/AS01E primary vaccination schedule) for the 5-17 months group; corresponding to Visit 5. The interim analysis concerned primary safety endpoints and the main secondary endpoints.

DETAILED DESCRIPTION:
The outcomes of interest (AESI, other AE leading to hospitalisation or death, and meningitis) as well as data on malaria morbidity and mortality were captured through active and enhanced hospitalisation surveillance in children less than (<) 5 years of age. Children enrolled in active surveillance were visited at their home at regular intervals during a period of 44 months. In addition to the home visits, all visits and hospitalisations to health care facilities were recorded during this period. Thereafter there was continuous monitoring of hospitalisations only; up to study end or up to the day the child reached 5 years of age, whichever occurred first. For all children enrolled in enhanced hospitalisation surveillance, all hospitalisation events were captured during the total study period. The protocol summary has been updated with protocol amendment 4 (dated 11-Dec-2015) information:

Rationale for amendment 3:

* Participant recruitment has been modified: approximately 20,000 children were to be enrolled in the active surveillance in the 6-12 weeks group (identified at first administration of DTP/HepB/Hib vaccine), to mimic administration of RTS,S/AS01E in the 6-12 weeks age group, and 20,000 children in the 5-17 months group (either selected children identified at first administration of DTP/HepB/Hib vaccine, or children aged 5 to <18 months and corresponding to a catch-up), to mimic administration of RTS,S/AS01E in the 5-17 months age group.
* The term "passive surveillance" has been replaced by the term "enhanced hospitalisation surveillance".
* The case definitions, ascertainment and laboratory investigation (including to determine aetiology) for meningitis cases have been clarified. The objectives and outcomes related to meningitis have been modified accordingly.
* Case ascertainment for AESI has been clarified.
* It was clarified that blood sampling was to be performed as per study procedures in case of AESI or meningitis. In case of neurological AESI or meningitis, if a cerebrospinal fluid (CSF) sample was taken as part of routine practice, part of the sample was stored. Only serious adverse events related to blood sampling were collected.
* Limitations due to the sample size and the study design have been further discussed.
* For clarity, consistency and comparability in the objectives, outcomes and methodologies, protocol amendment 3 text has been aligned in EPI-MALARIA-002 (115055) with the EPI-MALARIA-003 (115056) protocol.

Rationale for amendment 4:

* The background section has been updated with data about cerebral malaria from a post-hoc analysis of the Phase III study MALARIA-055.
* Additional secondary objectives have been added for estimation of probable meningitis and for estimation of the incidence of cerebral malaria using RDT and/or microscopy.
* The design and the analysis have been modified to take into account implementation of a 4th dose of RTS,S/AS01E. In addition, the follow-up period after the last dose has been extended to correspond to the follow-up period of the children enrolled in EPI-MAL-003 (i.e. 24 months after the 4th dose of RTS,S/AS01E). Indeed, home visits at 12 months and 24 months after the last RTS,S/AS01E dose will help to capture protocol-defined diseases that may have long risk window periods and that may not have been identified if the subject did not visit a health care facility, and to monitor the occurrence of malaria episodes for evaluation of vaccine effect. The age of the study population has been adapted accordingly (< 5 years).
* The section about sites participating to the study was updated following SAGE/MPAC recommendations of pilot implementations of RTS,S/AS01E in 3-5 distinct settings in SSA restricted to moderate-to-high transmission of malaria.
* The activities related to home visits to detect malaria cases, including training of community health workers for systematic measurement of body temperature of all children, and availability of malaria tests have been clarified for alignment with the EPI-MAL-003 protocol.
* It has been clarified that cases of malaria only detected during the annual visits planned for EPI-MAL-005 will not be included in the analysis of EPI-MAL-002. However, if the cases of malaria are detected during an EPI-MAL-005 home visit that coincides with a home visit scheduled in EPI-MAL-002, the events will be captured in EPI-MAL-002.
* The case definitions for malaria have been revised, according to the 3rd edition of the WHO guidelines for the treatment of malaria (2015). In addition, a case definition for cerebral malaria has been added.
* Case ascertainment by the external panel of experts has been clarified.
* It has been clarified that severe/cerebral malaria cases and other AE leading to hospitalisation or death were to be reviewed by the external panel of experts.
* The incidence of other AE leading to hospitalisation or death, meningitis and malaria morbidity and mortality were monitored in sub-populations of children with hemoglobinopathies and HIV-positive children.
* The section about analysis of co-primary objectives has been revised to mention that additional at risk periods were considered based on results as sensitivity analyses.
* The section about analysis of secondary objectives has been revised for clarification of potential variables that may be considered for models, in line with information collected in eCRF, and for estimation of the incidence of cerebral malaria.
* It has been clarified that an interim analysis was to be performed with the data collected on all subjects after 6 months of follow-up following the administration of dose 3 of DTP/HepB/Hib vaccine (6-12 weeks group), or 6 months after V3 (5-17 months group).
* The section about handling of missing data has been revised.
* It has been clarified that data about seasonal malaria chemoprevention was to be collected.

Other changes were made for simplification, clarification or consistency.

Rationale for amendment 5:

* In order to have a synergy with the WHO pilot implementation, the study size was reduced from 40,000 to 30,000 children in active surveillance with at least 20,000 children enrolled where the RTS,S/AS01E vaccine was implemented. Among the 30,000 children, approximately 15,000 children (with at least 10,000 children in sites where the vaccine was implemented) were to be enrolled in the 6-12 weeks group (to collect background data in this age group) and approximately 15,000 children (with at least 10,000 children in sites where the vaccine was implemented) were to be enrolled in the 5-17 months group (to mimic administration of RTS,S/AS01E in the 5-17 months age group). Study size updates involved multiple sections, e.g. Section 9.1 Study Design and Section 9.5 Study size.
* For multiple sections: the number of countries and number of study sites has been updated following the WHO announcement that the RTS,S/AS01E vaccine was first introduced in 3 countries (Ghana, Kenya and Malawi) through the MVIP.
* For multiple sections: estimation of the mortality rate, overall and by gender, has been added.
* For multiple sections: the informed consent process has been clarified "signed or witnessed and thumbprinted ICF".
* For multiple sections: "or equivalent surveillance system" has been added after Health and Demographic Surveillance System (HDSS) and the term "study site(s)" or "study area" has been added.
* For multiple sections: the replacement strategy has been updated.
* For multiple sections: the duration of the recruitment period has been removed, as it could/cannot be respected in all sites due to logistical constraints.
* For multiple sections: it was clarified that census rounds are scheduled at least once a year during the study periods instead of twice a year.
* The milestones in Section 6 have been updated.
* New sub-sections on "Severe malaria including cerebral malaria" and "Overall mortality by gender" have been added to Section 7.2 Safety results of the clinical development of RTS,S/AS01E.
* The wording of "secondary objectives" on "describe the causes of hospitalisation" and "estimate the incidence of cerebral malaria" has been changed, and the secondary objective "To describe the causes of death, overall and by gender" has been added in Section 8.2 and in the corresponding part of Section 4 Abstract.
* The opening paragraph of Section 8.2 Secondary Objectives and of the corresponding part of Section 4 Abstract has been updated.
* The wording of the last two "study variables" / "study endpoints" on "Occurrence of hospitalisations" and "Occurrence of death" has been modified in Section 9.3.2 and in the corresponding part of Section 4 Abstract.
* In Section 9.2.1 Study population: the text on "Estimated annual birth cohorts by study site" (Table 2) has been removed, with removal of planned number of sites in selected countries.
* Section 9.2.5.3 Meningitis has been edited, including addition of a new opening paragraph, addition of "turbid macroscopic aspect" as a sign of CSF abnormality, and clarification that clinically suspected meningitis cases included subjects with no CSF sample available and no alternative diagnosis.
* For consistency between the way the objectives and the endpoints were presented, and to avoid repeating several endpoints, the two sub-sections in Section 9.3.2 Secondary endpoints: "In children included in active or enhanced hospitalisation surveillance, prior to implementation of RTS,S/AS01E" and "In children included in active surveillance, prior to implementation of RTS,S/AS01E" have been replaced by one sub-section: "In children living in the study area, prior to implementation of RTS,S/AS01E", followed by all the secondary endpoints.
* In Section 9.4.3 Study EPI-MAL-005 "changes in environmental factors such as rainfall" has been added to the parameters assessed in EPI-MAL-005.
* Section 9.5 Study size has been updated as shown in bullet 1 above with greater detail on the estimates of observed incidence of events following dose administration based on either: 15,000 subjects, 10,000 subjects, the estimated birth cohort of 11,500 subjects and an estimated birth cohort of 17,250 children in Tables 6-9.
* Section 9.7.6 Analysis of secondary safety objectives has been updated, including analysis of cerebral malaria of the causes of death, overall and by gender.

Finally, changes in study personnel have been included on the protocol cover page

Rationale for amendment 6 Protocol Amendment 6 has been put in place to document that the EPI-MAL-002 study sites in Burkina Faso early terminated the study and that sites in Malawi, one of the countries where RTS,S/AS01E was introduced through the MVIP will not take part in the study.

GSK, in agreement with WHO, decided to terminate the study EPI-MAL-002 in the two sites located in Burkina Faso, i.e. Nouna and Sapone. Briefly, it was previously decided that Burkina Faso sites would continue participating in EPI-MAL-002 until study end. However, given that the MVIP will not be conducted in this country, there is no scientific value to collect additional data (the EPI-MAL-002 data collected in Burkina Faso will neither be used for the before-after analyses, nor for the generation of EPI-MAL-002 indicators that inform any other analyses of the EPI-MAL-003 study). Therefore, the study EPI-MAL-002 in Burkina Faso sites has been early terminated and data collected and recorded to date in those sites was to be reported in a descriptive way.

In order to align with the MVIP, the study sites for the GSK Phase IV studies have been selected from the 3 countries where the RTS,S/AS01E vaccine was implemented (Ghana, Kenya and Malawi). Considering the RTS,S/AS01E vaccine implementation date in Malawi was planned in October 2018, the baseline data that might be collected in Malawi in the EPI-MAL-002 study would be too limited to be relevant for the before/after comparisons in this country. Therefore, GSK, in agreement with the WHO, decided to focus the conduct of the EPI-MAL-002 study in Ghana and Kenya, not initiating the study in Malawi, and partially compensating the expected sample size from Malawi sites by using the high recruitment observed from sites in Kenya (Kombewa) and Ghana (Kintampo) and extending recruitment in Ghana (Navrongo), hence limiting the impact on the before/after comparison study power.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent provided from either the parent(s) or LAR of the subject.
* Subject living in the Health and Demographic Surveillance System (HDSS) area.
* For enrolment in active surveillance: children must be <18 months of age. OR
* For enrolment in enhanced hospitalisation surveillance: children must be <5 years of age and hospitalised at any time during the study.

Exclusion Criteria:

* Child in care.

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population was defined as those children living in the study areas who are < 5 years old.
Sampling Method: Non-Probability Sample
Enrollment: 36366 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Burkina Faso (2):
  - GSK Investigational Site, Ouagadougou
  - GSK Investigational Site, PO BOX 02 Nouna
- Ghana (2):
  - GSK Investigational Site, Kintampo
  - GSK Investigational Site, Navrongo
- GSK Investigational Site, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] RTS,S Epidemiology EPI-MAL-002 Study Group. Baseline incidence of meningitis, malaria, mortality and other health outcomes in infants and young sub-Saharan African children prior to the introduction of the RTS,S/AS01E malaria vaccine. Malar J. 2021 Apr 26;20(1):197. doi: 10.1186/s12936-021-03670-w. PMID 33902599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on 05 October 2015 in Burkina Faso site (which have early terminated the study and participants were not analysed), on 26 January 2016 in KE_Kombewa, on 07 February 2016 in GH_Kintampo and on 27 May 2017 in GH_Navrongo. Therefore, 26 January 2016 was considered the start date for the analysis.
Pre-assignment Details: Out of the 36366 participants initially enrolled in the study, 12939 participants from the Burkina Faso site were excluded from the According-To-Protocol (ATP) cohort. Therefore, 23427 participants formed the ATP cohort in Ghana and Kenya.
Period: Overall Study
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Started | 9032 | 9694 | 4701
Completed | 8060 | 8534 | 4218
Not Completed | 972 | 1160 | 483
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 91 | 110 | 4
Not completed — Lost to Follow-up | 168 | 194 | 138
Not completed — Death | 173 | 185 | 81
Not completed — Migrated from the study area | 538 | 648 | 181
Not completed — Enrollment in NCT03855995 study | 0 | 1 | 0
Not completed — Vaccination with RTS,S/AS01E vaccine | 2 | 0 | 0
Not completed — Other | 0 | 21 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance | Total
Number analyzed (Participants) | 9032 | 9694 | 4701 | 23427
Age, Continuous [Mean (Standard Deviation); unit: MONTHS] | 1.646 (0.2895) | 7.130 (5.1777) | 20.860 (15.4136) | 7.771 (10.3828)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4476 | 4754 | 2089 | 11319
  Male | 4556 | 4940 | 2612 | 12108
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Events of Specific Interest (AESI) From Month 0 to Month 79
Description: AESI were a predefined list of adverse events historically associated with vaccines other than RTS,S/AS01E or potentially associated with RTS,S/AS01E. This was because the RTS,S/AS01E vaccine contained new components not present in widely used vaccines at the time.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort, which included all evaluable participants who met all eligibility criteria, complied with the enrollment procedures defined in the protocol, and had no elimination criteria during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants | 12 | 11 | 16

2. Primary Outcome: Number of Participants With at Least One Adverse Event (AE) Leading to Hospitalization or Death From Month 0 to Month 79
Description: AEs assessed in children <5 years old, included in active or enhanced hospitalization surveillance, prior to implementation of RTS,S/AS01E.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: The analysis was performed on the ATP cohort, which included all evaluable participants who met all eligibility criteria, complied with the enrollment procedures defined in the protocol, and had no elimination criteria during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants | 1703 | 1763 | 4465

3. Primary Outcome: Number of Participants With at Least One Aetiology Confirmed Meningitis From Month 0 to Month 79
Description: Aetiology-confirmed meningitis was defined by the presence of symptoms and/or signs of meningitis and the identification of any known aetiologic agent (bacterial or not) in the Cerebrospinal Fluid (CSF).
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants | 1 | 1 | 11

4. Secondary Outcome: Number of Participants With at Least One Confirmed Meningitis Case From Month 0 to Month 79 (Final Classification)
Description: Final classification refers to the definitive categorization of meningitis cases after further investigation, typically involving additional laboratory testing and review by an external panel of experts. The criteria for final classification included:
  Aetiology-Confirmed Meningitis, which was defined if any known aetiologic agent (bacterial or not) was identified in the CSF sample.
  Probable Meningitis, which was defined if no aetiologic agent was identified in the CSF, but abnormalities were detected, or if there was a positive blood culture indicating bacterial infection.
  Clinically Suspected Meningitis, which was defined if all laboratory results were normal after second line laboratory testing, or if no CSF sample was available but no alternative diagnosis was found based on clinical symptoms and signs.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants
  Aetiology-confirmed and/or probable meningitis | 2 | 2 | 15
  Probable meningitis | 1 | 1 | 4
  Aetiology-confirmed, probable and/or clinically suspected meningitis | 3 | 7 | 24

5. Secondary Outcome: Number of Participants With at Least One Confirmed Meningitis Case Identified at Site Level From Month 0 to Month 79 (First Line Laboratory)
Description: First Line Laboratory refers to the initial laboratory testing conducted on cerebrospinal fluid (CSF) samples taken from patients suspected of having meningitis. The purpose of first line laboratory testing was to identify any bacterial agents present in the CSF or detect abnormalities that may indicate meningitis. The criteria for classifying cases at this stage included:
  Bacterial Confirmed Meningitis which was defined if a bacterial agent was identified in the CSF sample.
  Probable Meningitis which was defined if no bacterial agent was identified, but abnormalities were detected in the CSF or if there was a positive blood culture indicating bacterial infection.
  Clinically Suspected Meningitis which was defined if no bacterial agent was identified and all laboratory results were normal at the first line level, or if no CSF sample was available but no alternative diagnosis was found based on clinical symptoms and signs.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants
  Bacterial confirmed meningitis | 0 | 1 | 3
  Probable meningitis | 5 | 5 | 23
  Clinically suspected meningitis | 4 | 8 | 13

6. Secondary Outcome: Number of Participants With Risk Factors for AESI, Meningitis and Malaria Among Hospitalized Participants
Description: As per Statistical analysis plan, Univariate and multivariate Poisson regression models for analysis of potential risk factors for AESI, aetiology-confirmed meningitis and cerebral malaria were only planned to be conducted if there were a minimum of 10 cases.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: The analysis was planned to perform on ATP cohort, which included all evaluable participants who met all eligibility criteria, complied with enrollment procedures defined in protocol, and had no elimination criteria during study. As per analysis plan, Poisson regression models for analyzing potential risk factors for AESI, aetiology-confirmed meningitis, cerebral malaria, and death were only planned if there were at least 10 cases. Since the case count was below 10, no analysis was conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants | NA [NA to NA] — As per Statistical analysis plan, Univariate and multivariate Poisson regression models for analysis of potential risk factors for AESI, aetiology-confirmed meningitis, cerebral malaria and death were only planned to be conducted if there were a minimum of 10 cases. Since the number of cases were less than 10, analysis was not performed. | NA [NA to NA] — As per Statistical analysis plan, Univariate and multivariate Poisson regression models for analysis of potential risk factors for AESI, aetiology-confirmed meningitis, cerebral malaria and death were only planned to be conducted if there were a minimum of 10 cases. Since the number of cases were less than 10, analysis was not performed. | NA [NA to NA] — As per Statistical analysis plan, Univariate and multivariate Poisson regression models for analysis of potential risk factors for AESI, aetiology-confirmed meningitis, cerebral malaria and death were only planned to be conducted if there were a minimum of 10 cases. Since the number of cases were less than 10, analysis was not performed.

7. Secondary Outcome: Incidence Rates of Death After the Virtual Secondary Schedule (Secondary Dose of DTP/HepB/Hib Administered at Day 31) for the Active Surveillance 6-12 Weeks and Active Surveillance 5-17 Weeks Groups
Description: Incidence rate was calculated by dividing the number of participants reporting at least one event over the follow-up period by the total person-time. Analysis of this outcome measure were reported only for the Active surveillance 6-12 weeks and Active surveillance 5-17 months groups, as the participants in the Enhanced hospitalization surveillance group were not administered with the DTP/HepB/Hib vaccine.
Time Frame: Day 31 to approximately Month 13 (Within an at-risk period of 12 months after virtual secondary schedule)
Population: The analysis was performed only on the participants from the Active surveillance 6-12 weeks and Active surveillance 5-17 months groups, as only they received a secondary dose of DTP/HepB/Hib administered at Day 31. The participants belonged to the ATP cohort, met all eligibility criteria, complied with the enrollment procedures defined in the protocol and had no elimination criteria during the study.
Measure: Number (95% Confidence Interval); unit: events per 100,000 person-years
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months
Number analyzed (Participants) | 8871 | 9339
events per 100,000 person-years | 677.42 [560.72 to 811.25] | 642.97 [531.30 to 771.18]

8. Secondary Outcome: Number of Participants Hospitalized With Causes (Including Those Attributed to an AESI, Other AE, Meningitis, or Malaria) From Month 0 to Month 79
Description: Hospitalized cases attributed to an AESI, other AE, meningitis, or malaria were assessed in children <5 years old, included in active or enhanced hospitalization surveillance, prior to implementation of RTS,S/AS01E.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants
  Hospitalization - AESI | 12 | 11 | 16
  Hospitalization - Other AE | 1703 | 1763 | 4465
  Hospitalization - Meningitis | 3 | 7 | 24
  Hospitalization - Malaria | 1013 | 1224 | 2458
  Hospitalization - P. falciparum | 1007 | 1218 | 2068

9. Secondary Outcome: Number of Participants Reported Deaths From Month 0 to Month 79
Description: Mortality events were assessed in children <5 years old, included in active or enhanced hospitalization surveillance, prior to implementation of RTS,S/AS01E.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants | 173 | 183 | 80

10. Secondary Outcome: Number of Participants With Malaria Cases Reported Using Rapid Diagnostic Test (RDT) and/or Microscopy From Month 0 to Month 79
Description: Any malaria includes uncomplicated and severe cases, including cerebral malaria. Uncomplicated is defined as: Plasmodium parasitaemia greater than (>) 0 detected by microscopy and/or RDT, fever (temperature ≥ 37.5°C) and no signs of severity or evidence (clinical or laboratory) of vital organ dysfunction. Severe is defined as: P. falciparum parasitaemia > 0 detected by microscopy and/or RDT and one or more of the following: impaired consciousness, prostration, multiple convulsions, acidosis, hypoglycaemia, severe malarial anaemia, renal impairment, jaundice, pulmonary oedema, significant bleeding, shock, hyperparasitaemia. Cerebral malaria is defined as severe P. falciparum malaria with impaired consciousness.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants
  Any Malaria | 5072 | 5714 | 2458
  Severe Malaria | 202 | 247 | 550
  Cerebral Malaria cases | 8 | 9 | 20

11. Secondary Outcome: Number of Participants With All Anaemia and Severe Anaemia Cases Among Hospitalized Children From Month 0 to Month 79
Description: Cases of anaemia were defined as follow: All anaemia: haemoglobin lower than 11grams per deciliter (g/dL). Severe anaemia: haemoglobin lower than 7g/dL .
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants
  All anaemia | 1132 | 1215 | 2783
  Severe anaemia | 254 | 338 | 758

12. Secondary Outcome: Number of Participants With All Cause Hospitalizations and Hospitalizations Attributed to Malaria (Including P. Falciparum) From Month 0 to Month 79
Description: The hospitalization cases were assessed in children <5 years old, included in active surveillance, prior to implementation of RTS,S/AS01E. Hospitalisation for malaria (including P. falciparum) was defined as a hospitalized participants with malaria (including P. falciparum malaria) and for whom malaria is the primary cause of hospitalization.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants
  Hospitalisation - All causes | 1788 | 1907 | 4701
  Hospitalisation - P. falciparum | 1007 | 1218 | 2441

13. Secondary Outcome: Number of Participants Reported All-cause Mortality and Deaths Attributed to Malaria (Overall and by Gender) From Month 0 to Month 79
Description: All cause mortality and death attributed to malaria are summarized by overall and gender.
Time Frame: During the entire study period (From Month 0 up to Month 79)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
Number analyzed (Participants) | 9032 | 9694 | 4701
Participants
  Death- All cause(Male) | 81 | 105 | 49
  Death- All cause(Female) | 92 | 78 | 31
  Death(Overall) | 173 | 183 | 80
  Death - Malaria(Male) | 18 | 34 | 0
  Death - Malaria(Female) | 24 | 21 | 1
  Death - Malaria(Overall) | 42 | 55 | 1

ADVERSE EVENTS:
Time Frame: From Day 1 to Month 79
Description: SAEs were recorded as as a result of the blood draw for a suspected AESI or meningitis. Death related to study procedure were only considered as SAEs. Solicited and -Unsolicited adverse events(Non-Serious adverse events) were not collected since the capillary blood sampling was the only invasive procedure involved in this study.
Arm/Group | Active Surveillance 6-12 Weeks | Active Surveillance 5-17 Months | Enhanced Hospitalization Surveillance
All-Cause Mortality (participants affected / at risk) | 173/9032 | 183/9694 | 80/4701
Serious Adverse Events (participants affected / at risk) | 0/9032 | 0/9694 | 0/4701
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study limitations included influences on case detection and ascertainment due to factors such as medical supply shortages, limited investigational capacities, and reduced availability of medical personnel during strikes and elections. Despite efforts to improve case detection, a "study effect" could still be anticipated. Modifications in malaria case definition and occasional missed home visits for a small number of participants might have had a minimal impact on interpretation of study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinic.

DOCUMENTS (2):
  • Study Protocol (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT02374450/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT02374450/SAP_001.pdf